CLINICAL TRIAL: NCT03318978
Title: Benzo[a]Pyrene Ultralow Dose-Response Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); Lawrence Livermore National Laboratory (Other); Pacific Northwest National Laboratory (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Williams, Helen P. Rumbel Professor for Cancer Prevention, Oregon State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LPI-8233; R01ES028600 (NIH)
Record Dates: First submitted 2017-10-17; First posted 2017-10-24 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Environmental Exposure
Keywords: Benzo[a]pyrene; Accelerator Mass Spectrometry; Polycyclic Aromatic Hydrocarbons

STUDY DESIGN:
Masking Description: Deidentified samples will be analyzed by AMS at Lawrence Livermore National Laboratory and the pharmacokinetics determine at Pacific Northwest National Laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 25 ng dose, 50 ng dose, 100 ng dose, 250 ng dose (Experimental): Cycle 1: Capsule containing 25 ng (2.7 nCi) [14C]-benzo[a]pyrene (BaP).
  Cycle 2: Capsule containing 50 ng (2.7 nCi) [14C]-benzo[a]pyrene (BaP).
  Cycle 3: Capsule containing 100 ng (2.7 nCi) [14C]-benzo[a]pyrene (BaP).
  Cycle 4: Capsule containing 250 ng (2.7 nCi) [14C]-benzo[a]pyrene (BaP).
  At least 3 weeks will pass between cycles as a washout period.
  Interventions: Drug: [14C]-benzo[a]pyrene

INTERVENTIONS:
Drug: [14C]-benzo[a]pyrene — Oral micro-dose range (25, 50, 100 and 250 ng)
  Other Names: Carcinogenic PAH environmental pollutant

SUMMARY:
Evaluation of the pharmacokinetics for [14C]-benzo[a]pyrene ([14C]-BaP) and metabolites in plasma and urine over 48 hours following 4 oral doses of 25, 50, 10 and 250 ng (2.7-27 nCi).

DETAILED DESCRIPTION:
The pharmacokinetics for [14C]-BaP and metabolites will be assessed by UHLPC-Accelerator Mass Spectrometry (AMS, Lawrence Livermore National Laboratory) in plasma and urine collected over 48 hours following oral doses of 25, 50, 100 or 250 ng (2.7-27 nCi). Metabolite profiles and kinetics of elimination over this dose range are predicted to be consistent with a BaP physiologically based pharmacokinetic (PBPK) model developed by Pacific Northwest National Laboratory (PNNL). A non-smoker, not exposed occupationally, receives 270-700 ng of BaP daily; about 95% dietary. The WHO has set an estimated safe daily lifetime (70 year/70 Kg individual, cancer endpoint) exposure to BaP of 42-350 ng. This protocol represents de minimus risk.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for women:

  * Age 21-65 (inclusive)
  * Must be post-menopausal or have had surgical sterilization to eliminate any possibility for fetal exposure
  * Willing to defer blood donation for one month before, throughout, and one month after completion of study activities
  * Willing to avoid consuming cruciferous vegetables, I3C or DIM supplements, smoked or cured meat or cheeses, or charcoal-grilled meats for 2 weeks prior to and during each study cycle (gas grilled foods acceptable)

Inclusion criteria for men:

* Age 21-65 (inclusive)
* Willing to defer blood donation for one month before, throughout, and one month after completion of study activities
* Willing to avoid consuming cruciferous vegetables, I3C or DIM supplements, smoked or cured meat or cheeses, or charcoal-grilled meats for 2 weeks prior to and during each study cycle (gas grilled foods acceptable)

Exclusion Criteria:

Exclusion criteria for both men and women:

* Smoker (tobacco or other substances) or use of smokeless tobacco in past 3 months or living with smoker
* Regular use of medications that affect gut motility or nutrient absorption (e.g. cholestyramine, sucralfate, orlistat, pro- or anti-motility agents)
* History of gastrointestinal surgery (e.g. bariatric surgery, cholecystectomy) or gastrointestinal disorder (Crohn's disease, celiac disease, IBS, or colitis)
* Current or history of kidney or liver disease
* Prior high-dose 14C exposure from medical tests. (micro-dose 14C exposure not exclusionary)
* Occupational PAH exposure (e.g. roofers, asphalt pavers, fire-fighters, etc.)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Facility, 407 Linus Pauling Science Center, Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified samples sent to Lawrence Livermore National Laboratory Deidentified data sent to Pacific Northwest National Laboratory

RESULTS

PARTICIPANT FLOW:
Groups:
- 25 ng Dose, 50 ng Dose, 100 ng Dose, 250 ng Dose: [14C]-benzo[a]pyrene: Oral micro-dose range (25, 50, 100 and 250 ng)
  At least 3 weeks must pass between each capsule dose administration.
Period: Overall Study
Arm/Group | 25 ng Dose, 50 ng Dose, 100 ng Dose, 250 ng Dose
Started | 8 (One participant consented to participate and voluntarily withdrew prior to beginning the study protocol (no BaP doses administered).)
Completed | 7
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | 25 ng Dose, 50 ng Dose, 100 ng Dose, 250 ng Dose
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration Cmax
Description: Determination of highest concentration in plasma. Blood samples collected at 0 (baseline), 0.25, 0.5, 1, 2, 3, 4, 8, 24, and 48 hour after dosing. All time points were used to determine peak plasma concentration Cmax.
Time Frame: 0-48 hours for each of the 4 dosing cycles with a washout period of 3 weeks between each dosing cycle
Measure: Mean (Standard Deviation); unit: fg [14C]-BaP/mL plasma
Groups:
- 25 ng, 50 ng, 100 ng, and 250 ng Doses: Cycle 1: Capsule containing 25 ng [14C]-benzo[a]pyrene (BaP).
  Cycle 2: Capsule containing 50 ng [14C]-benzo[a]pyrene (BaP)
  Cycle 3: Capsule containing 100 ng [14C]-benzo[a]pyrene (BaP)
  Cycle 4: Capsule containing 250 ng [14C]-benzo[a]pyrene (BaP)
  At least 3 weeks will pass between cycles as a washout period.
Arm/Group | 25 ng, 50 ng, 100 ng, and 250 ng Doses
Number analyzed (Participants) | 7
fg [14C]-BaP/mL plasma
  25 ng [14C]-BaP | 2.51 (2.53)
  50 ng [14C]-BaP | 5.68 (4.70)
  100 ng [14C]-BaP | 13.8 (9.52)
  250 ng [14C]-BaP | 8.99 (7.08)

2. Secondary Outcome: Time at Highest Plasma Concentration Tmax
Description: Determination of time at which plasma concentration is highest. Blood samples collected at 0 (baseline), 0.25, 0.5, 1, 2, 3, 4, 8, 24, and 48 hour after dosing. All time points were used to determine Tmax, time at highest plasma concentration.
Time Frame: 0-48 hours for each of the 4 dosing cycles with a washout period of 3 weeks between each dosing cycle
Measure: Median (Full Range); unit: hour
Groups:
- 25 ng Dose, 50 ng Dose, 100 ng Dose, 250 ng Dose: Cycle 1: Capsule containing 25 ng (2.7 nCi) [14C]-benzo[a]pyrene (BaP).
  Cycle 2: Capsule containing 50 ng (2.7 nCi) [14C]-benzo[a]pyrene (BaP).
  Cycle 3: Capsule containing 100 ng (2.7 nCi) [14C]-benzo[a]pyrene (BaP).
  Cycle 4: Capsule containing 250 ng (2.7 nCi) [14C]-benzo[a]pyrene (BaP).
  At least 3 weeks will pass between cycles as a washout period.
  [14C]-benzo[a]pyrene: Oral micro-dose range (25, 50, 100 and 250 ng)
Arm/Group | 25 ng Dose, 50 ng Dose, 100 ng Dose, 250 ng Dose
Number analyzed (Participants) | 7
hour
  25 ng [14C]-BaP | 0.5 [0.5 to 4.0]
  50 ng [14C]-BaP | 0.5 [0.5 to 1.0]
  100 ng [14C]-BaP | 0.5 [0.5 to 1.0]
  250 ng [14C]-BaP | 0.5 [0.5 to 3.0]

3. Secondary Outcome: Area Under Plasma Concentration Versus Time Curve AUC
Description: Integration of concentration over time. Blood samples collected at 0 (baseline), 0.25, 0.5, 1, 2, 3, 4, 8, 24, and 48 hour after dosing. All time points were used to determine AUC.
Time Frame: 0-48 hours for each of the 4 dosing cycles with a washout period of 3 weeks between each dosing cycle
Measure: Mean (Standard Deviation); unit: fg [14C]-BaP/mL plasma x hour
Arm/Group | 25 ng Dose, 50 ng Dose, 100 ng Dose, 250 ng Dose
Number analyzed (Participants) | 7
fg [14C]-BaP/mL plasma x hour
  25 ng [14C]-BaP | 12.2 (14.5)
  50 ng [14C]-BaP | 19.6 (15.7)
  100 ng [14C]-BaP | 88.5 (14.1)
  250 ng [14C]-BaP | 68.6 (60.4)

4. Secondary Outcome: Rate of Elimination (k1e)
Description: Determination of constants for rate of elimination from plasma. Blood samples collected at 0 (baseline), 0.25, 0.5, 1, 2, 3, 4, 8, 24, and 48 hour after dosing. All time points were used to determine k1e.
Time Frame: 0-48 hours for each of the 4 dosing cycles with a washout period of 3 weeks between each dosing cycle
Measure: Mean (Standard Deviation); unit: hour(-1)
Arm/Group | 25 ng Dose, 50 ng Dose, 100 ng Dose, 250 ng Dose
Number analyzed (Participants) | 7
hour(-1)
  25 ng [14C]-BaP | 12.2 (14.5)
  50 ng [14C]-BaP | 19.6 (15.7)
  100 ng [14C]-BaP | 88.5 (14.1)
  250 ng [14C]-BaP | 68.6 (64.0)

ADVERSE EVENTS:
Time Frame: 48.5 hours for each of 4 dosing cycles with a 3-week washout period between each dosing cycle. Participants were assessed for adverse events 15 minutes prior to the [14c]-BaP dose administration (time= 0 hour) until 15 minutes after the final blood sample collection time point (time = 48 hour) and removal of the peripheral IV catheter.
Description: The definitions of adverse event and serious adverse event used to determine incidence are consistent with clinicaltrials.gov definitions. Each participant was verbally asked about the occurrence of adverse events at each clinical visit by the research nurse.
Arm/Group | 25 ng Dose, 50 ng Dose, 100 ng Dose, 250 ng Dose
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT03318978/Prot_SAP_ICF_000.pdf